CLINICAL TRIAL: NCT01430975
Title: A Prospective Study to Estimate Inadvertent Radiation Exposure From Strontium Isotopes in Patients Who Have Undergone CardioGen-82® PET MPI Scanning at Two Clinical Sites
Brief Title: Prospective Evaluation of Strontium in Patients After CardioGen-82 PET MPI Scanning at Two Clinical Sites
Status: Completed | Type: Observational
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CGEN-104
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Radiation Exposure
Keywords: Radiation Exposure; Rubidium 82; Strontium 82; Strontium 85

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CardioGen-82 — CardioGen-82 was not administered as part of this trial but the patients enrolled had to have received CardioGen-82 previously
Drug: CardioGen-82 — Patients do not received CardioGen-82 as part of this study. To be in the study they would have had to receive CardioGen-82 previously.

SUMMARY:
This study is to be performed at two clinical sites where patients received CardioGen-82 during the time period January to June, 2011 and where patients were scanned chronologically near to the index patients (2 days before or after). Of these, it is planned that at least 30 patients will be entered in this trial. Index patient is the term applied to individuals who had radiation spectra indicative of Sr-82 and Sr-85 detected by hand-held survey meters.

DETAILED DESCRIPTION:
This clinical study protocol will use a three tier approach consisting of the following examinations:

* Patient examination with Survey Meter: The patient will first be tested at the clinical sites using a survey meter. In those patients whose radiation count is ≥ 2 times above background count using a standard survey meter, the presence of Sr-82 and/or Sr-85 will be assessed through a quantitative reading from a calibrated portable isotope identifier.
* Patient examination with Portable Isotope Identifier: This examination will be done by use of a portable isotope identifier, which will be supplied by the Sponsor to the study sites. An assessor, independent to the study site and will perform the examination. In those patients whose radiation count is ≥ 2 times above background count using a standard survey meter, the presence of Sr-82 and/or Sr-85 will be assessed through a quantitative reading from a calibrated portable isotope identifier. The reading will be forwarded along with the date of the reading, the date of the patient's CardioGen-82® scan, and the total dose of CardioGen-82® administered to the patient, to an independent medical expert, independent to the study site, who will back-calculate an estimated dose of Sr-82 and/or Sr-85 from these data.
* Patient examination at Oak Ridge National Laboratory: Any patient whose estimated dose of Sr-82 exceeds the specified limit of 0.02 microcuries per mCi Rb-82 administered, and/or whose estimated dose of Sr-85 exceeds the specified limit of 0.2 microcuries per mCi Rb-82 administered, will be asked to travel to Oak Ridge National Laboratory in Tennessee, for accurate whole body scanning. Scan data from Oak Ridge National Laboratories will be analyzed by one or more independent medical experts to accurately back-calculate exposure to Sr-82 and/or Sr-85, and to estimate health hazard for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Gave informed consent to participate in the study;
* Received CardioGen-82 that has been eluted from the generator in close proximity (2 days before or after) the index patients.

Exclusion Criteria:

-Any patient previously enrolled in and completed this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population would come from the two sites who administered CardioGen-82® to the index patients. Each site that agrees to participate will enroll patients administered CardioGen-82 2 days before and 2 days after the use of that generator.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Determination of radiation exposure from Sr-82 and/or Sr-85 | on average within 24 hours
  To determine radiation exposure from Sr-82 and/or Sr-85 in patients administered CardioGen-82® for PET MPI at the two sites reporting Sr-82/Sr-85 breakthrough
Determination of extent of SR-82/Sr-85 exposure, if positive exposure is detected | within 2 weeks
  To determine the extent of the Sr-82/Sr-85 exposure, in the subset of patients with positive testing exceeding the specified threshold for the breakthrough of Sr-82/Sr-85, by performing whole body scanning at Oak Ridge National Laboratory for eventual health hazard assessment

CONTACTS AND LOCATIONS:
Overall Officials: Steven Sireci, M.D., Study Director — Bracco Diagnostics, Inc
Locations (1):
- Bracco Diagnostics, Inc., Princeton, New Jersey, United States